CLINICAL TRIAL: NCT04946084
Title: Dynamic Change and Immune Response to Nasopharyngeal Carriage and Acute Otitis Media Pathogens
Acronym: AOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Michael Pichichero, Director, Rochester General Hospital Research Institute, Rochester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 2031 A
Record Dates: First submitted 2021-05-24; First posted 2021-06-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Tympanocentesis; Therapeutic Irrigation; Nasal Lavage; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Children (Other): Samples taken from nasal swabs, nasal wash, blood draws and in the case of acute otitis media, tympanocentesis
  Interventions: Procedure: Tympanocentesis; Other: Nasal Phalangeal Swab and Wash; Other: Blood Draw

INTERVENTIONS:
Procedure: Tympanocentesis — When acute otitis media is diagnosed, local anesthetic applied, small hole placed in eardrum, middle ear fluid extracted.
  Other Names: Ear Tap
Other: Nasal Phalangeal Swab and Wash — Nasal phalangeal swab used to retrieve sample. Nasal wash used to retrieve sample.
  Other Names: Nasal Swab, Nasal Wash
Other: Blood Draw — Venipuncture

SUMMARY:
The investigators seek to conduct a prospective, longitudinal study to identify the dynamic changes in nasopharyngeal (NP) colonization patterns and acute otitis media (AOM) etiology involving antibiotic-resistant Streptococcus pneumoniae (Spn) and Haemophilus influenzae (Hflu).

DETAILED DESCRIPTION:
The investigator's proposed study design involves 2 cohorts. Cohort 1: Collection of middle ear fluid(MEF), NP samples and blood at onset of AOM from otitis prone children and those who have AOM antibiotic treatment failure since these children more frequently harbor antibiotic resistant strains. Children will then be followed prospectively thereafter, collecting NP samples at pre-determined time points when the children are healthy (see cohort 2) and MEF, NP samples and blood if subsequent AOM infections occur. Cohort 2: Healthy children from whom we will prospectively collect NP samplings and blood at any of 7 pre-determined time points (age 6, 9, 12, 15, 18, 24, and/or 30-36 months old as they occur within the study time-frame) to assess commensal carriage of Spn and Hflu. MEF will be obtained from the participants at any AOM occurring, including the first and any subsequent AOM infection. Concurrently detailed demographic, vaccination, epidemiologic and risk factor data known to influence AOM epidemiology will be collected, providing scientific rigor.

Viral respiratory infections will be another focus during this project. The investigators will characterize dynamic changes in patterns of viral co-infections at onset of AOM including the common respiratory viruses RSV A, B, influenza A, B, parainfluenzae virus type 3, rhinovirus, enterovirus, human metapneumovirus, human bocavirus, adenovirus B, C and SARS-CoV-2. The studies will involve viral identification, evaluation of viral/bacterial (otopathogen) interactions and mucosal and systemic immune responses.

The investigators have identified multiple deficiencies in innate and adaptive immunity among young children who are AOM prone and introduced the term "prolonged neonatal-like immune profile (PNIP) because of striking similarities that resemble neonatal immunity. Another focus of this project will be to expand understanding of the central immune deficiencies of APM prone children using blood samples.

A a serum correlate of protection has been defined to predict the effectiveness of pneumococcal conjugate vaccines using blood samples linked to occurrence of NP colonization and AOM events in recent past work. Blood will be used to continue this work.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject age 6 to 12 months + 30 days at the time of enrollment when healthy or up to 36 months old + 30 days with an ear infection.
* Subject has received full (3 dose) infant series of PCV.
* Parent/legal guardian must be able and willing to bring subject to all study visits

Exclusion Criteria:

* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in the study.
* Participation in another investigational or interventional trial within the 28-day period before enrollment and during the conduct of the study. Participation in observational studies is permitted.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize which bacterial strains in the NP | 30 months
  Identify the presence of Streptococcus pneumoniae, Haemophilus influenzae and Moraxella catharralis in the nasopharynx of children using in vitro culture

SECONDARY OUTCOMES:
Characterize which bacterial strains are AOM causing pathogens | 30 months
  Identify the presence of Streptococcus pneumoniae, Haemophilus influenzae and Moraxella catharralis in the nasopharynx of children using in vitro culture

OTHER OUTCOMES:
Characterize dynamic changes in patterns of viral co-infections at onset of AOM | 30 months
  Identify respiratory viruses present in the nasopharynx at onset of acute otitis media in young children using polymerase chain reaction methods.
Determine immune responses after NP carriage and AOM infections by the common bacterial respiratory pathogens. | 30 Months
  Measure serum and nasopharyngeal antibody levels to common bacterial and viral respiratory pathogens with ELISA and immune cellular responses (B cells, T cells, Antigen Presenting cells using flow cytometry and ELISPOT
Determine the serum antibody response that correlates with protection against NP colonization and AOM. | 30 months
  Establish a correlate of protection for pneumococcal serotypes that colonize the nasopharynx and cause acute otitis media in young children using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pichichero, MD, Principal Investigator — Rochester General Hospital Research Institute
Locations (1):
- Rochester General Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No